CLINICAL TRIAL: NCT01014143
Title: Evaluating Commercial Anti-Plaque Products and Oral Rinse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2007-PLA-15-RR
Record Dates: First submitted 2008-09-26; First posted 2009-11-16 (Estimated); Results first posted 2009-11-16 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Fluorides; chlorhexidine gluconate; Triclosan; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluoride toothpaste (Placebo Comparator): Negative control
  Interventions: Drug: Fluoride
- Triclosan/Fluoride toothpaste (Active Comparator): positive control toothpaste
  Interventions: Drug: Fluoride, triclosan
- Chlorhexidine Oral Rinse (Active Comparator): Positive Control mouthrinse
  Interventions: Drug: Chlorhexidine digluconate

INTERVENTIONS:
Drug: Fluoride — Half mouth toothbrushing twice a day for four days.
  Other Names: fluoride toothpaste
  Arms: Fluoride toothpaste
Drug: Chlorhexidine digluconate — Mouth rinsing with 15 ml for 30 seconds twice a day for four days.
  Other Names: Periogard oral rinse
  Arms: Chlorhexidine Oral Rinse
Drug: Fluoride, triclosan — Half mouth Brushing twice daily
  Other Names: Total toothpaste
  Arms: Triclosan/Fluoride toothpaste

SUMMARY:
Clinical research study to determine the anti-plaque efficacy of commerical dentifrices and an oral rinse.

DETAILED DESCRIPTION:
This clinical research study was to train new examiners for short term plaque clinical methodologies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers at least 18 years of age.
* Good general health.
* Must sign informed consent form.
* Minimum of 20 natural uncrowned teeth (excluding third molars) must be present.
* No history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study.

Exclusion Criteria:

* Subjects unable or unwilling to sign the informed consent form.
* Medical condition which requires pre-medication prior to dental visits/procedures.
* Moderate or advanced periodontal disease or heavy dental tartar (calculus).
* Two or more decayed untreated dental sites at screening.
* Other disease of the hard or soft oral tissues.
* Impaired salivary function (e.g. Sjogren's syndrome or head and neck irradiation).
* Use of medications that are currently affect salivary function.
* Use of antibiotics or antimicrobial drugs within 30 days prior to study visit #1.
* Allergy to chlorhexidine.
* Pregnant or nursing women.
* Participation in any other clinical study within 1 week prior to enrollment into this study.
* Use of tobacco products.
* Subjects who must receive dental treatment during the study dates.
* Current use of Antibiotics for pre-medication for dental treatment or for any other purpose.
* Presence of an orthodontic appliance that interferes with plaque scoring.
* History of allergy to common dentifrice ingredients.
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy).

Ages: 23 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cronin, DDS, Principal Investigator
Locations (1):
- New Institutional Service Company, Northfield, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed by the clinical site
Groups:
- Fluoride Toothpaste First: Fluoride first, 1 week washout,triclosan/fluoride (Total) second,1 week washout, Oral Rinse last
- Total Toothpaste First: triclosan/fluoride (Total)toothpaste first,1 week washout, Chlorhexidine rinse second, 1 week washout and fluoride toothpaste last
- Chlorhexidine Oral Rinse First: chlorhexidine oral rinse first,1 week washout, fluoride toothpaste second, 1 week washout, triclosan/fluoride (Total)last
Period: First Intervention
Arm/Group | Fluoride Toothpaste First | Total Toothpaste First | Chlorhexidine Oral Rinse First
Started | 10 | 9 | 9
Completed | 10 | 9 | 9
Not Completed | 0 | 0 | 0
Period: Washout Period After 1st Intervention
Arm/Group | Fluoride Toothpaste First | Total Toothpaste First | Chlorhexidine Oral Rinse First
Started | 10 | 9 | 9
Completed | 10 | 9 | 9
Not Completed | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Fluoride Toothpaste First | Total Toothpaste First | Chlorhexidine Oral Rinse First
Started | 10 | 9 | 9
Completed | 8 | 9 | 9
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Period: Washout After 2nd Intervention
Arm/Group | Fluoride Toothpaste First | Total Toothpaste First | Chlorhexidine Oral Rinse First
Started | 8 | 9 | 9
Completed | 8 | 9 | 9
Not Completed | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Fluoride Toothpaste First | Total Toothpaste First | Chlorhexidine Oral Rinse First
Started | 8 | 9 | 9
Completed | 8 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Toothpaste: triclosan/fluoride toothpaste (positive control toothpaste)
- Chlorhexidine Oral Rinse: chlorhexidine mouthrinse (positive control rinse)
- Total: Total of all reporting groups
Arm/Group | Fluoride Toothpaste | Total Toothpaste | Chlorhexidine Oral Rinse | Total
Number analyzed (Participants) | 10 | 9 | 9 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 9 | 28
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.6 (15.1) | 39 (9.2) | 47.2 (9.6) | 44.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 9 | 22
  Male | 3 | 3 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 9 | 28

OUTCOME MEASURES:

1. Primary Outcome: Plaque Index
Description: Plaque scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque,3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Time Frame: Four days
Population: per protocol. 2 subjects missed appointments and did not complete two of the study treatment periods.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fluoride Toothpaste | Total Toothpaste | Chlorhexidine Oral Rinse
Number analyzed (Participants) | 28 | 26 | 26
Units on a scale | 2.63 (0.61) | 2.65 (0.56) | 1.23 (0.59)
Statistical Analysis 1: Comparison: Fluoride Toothpaste vs Total Toothpaste vs Chlorhexidine Oral Rinse; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: subjects were examined at each clinic visit for any signs of side effects while using the study products. If any subject developed any potential side effect while using the study products, they called 24 hour contact number to report it and made an appointment with the clinician to have the side effect evaluated.
Arm/Group | Fluoride Toothpaste First | Total Toothpaste First | Chlorhexidine Oral Rinse First
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 1/28 | 1/28 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Fluoride Toothpaste First (N=28) | Total Toothpaste First (N=28) | Chlorhexidine Oral Rinse First (N=28)
Upset stomach - non related to product use (Social circumstances) | 1/26 (1) | 0/26 (0) | 0/26 (0) — All events resolved in the same day to 3 days after reporting. Adverse events reported in this study were determined not to be related to study product use.
Sinus headache - non related to product use (Social circumstances) | 0/26 (0) | 1/26 (1) | 0/26 (0) — All events resolved in the same day to 3 days after reporting. Adverse events reported in this study were determined not to be related to study product use.
Menstrual cramps (Social circumstances) | 0/26 (0) | 0/26 (0) | 1/26 (1) — All events resolved in the same day to 3 days after reporting. Adverse events reported in this study were determined not to be related to study product use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days